CLINICAL TRIAL: NCT05142631
Title: Single Center, Open, Single Arm Phase II Clinical Study of Fruquintinib in the Treatment of Soft Tissue Sarcoma
Brief Title: Fruquintinib in the Treatment of Soft Tissue Sarcoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-013-CH05 IIT-STS
Record Dates: First submitted 2021-11-21; First posted 2021-12-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Soft Tissue Sarcoma
Keywords: soft tissue sarcoma; Fruquintinib
MeSH Terms: conditions — Sarcoma | interventions — HMPL-013

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fruquintinib in soft tissue sarcoma (Experimental): Fruquintinib : 5mg, once a day (QD), oral on an empty stomach or after a meal, taken with 100 ~ 200ml drinking water for 3 weeks and stopped for 1 week.
  Interventions: Drug: Fruquintinib

INTERVENTIONS:
Drug: Fruquintinib — To observe the efficacy and safety of Fruquintinib in the first-line treatment of desmoplastic small round cell tumor, epithelioid hemangioendothelioma, solitary fibroma or second-line and posterior line treatment of angiosarcoma.

SUMMARY:
To evaluate the efficacy of Fruquintinib in patients with chemotherapy insensitive or chemotherapy resistant soft tissue sarcoma

DETAILED DESCRIPTION:
This trial is an open, single arm, single center, prospective phase II clinical study. Objective:To observe the efficacy and safety of Fruquintinib in the first-line treatment of desmoplastic small round cell tumor, epithelioid hemangioendothelioma, solitary fibroma or second-line and posterior line treatment of angiosarcoma.

ELIGIBILITY:
Inclusion Criteria:

Only those who meet all of the following criteria can be selected:

1. Fully understand this study and voluntarily sign the informed consent form;
2. Male or female subjects / patients aged ≥ 18 years;
3. Non operative desmoplastic small round cell tumor, epithelioid hemangioendothelioma, solitary fibroma and angiosarcoma with failed chemotherapy confirmed by histopathology;
4. Patients with desmoplastic small round cell tumor, epithelioid hemangioendothelioma, solitary fibroma or angiosarcoma who failed to receive anti angiogenesis drugs in the past.
5. At least one measurable lesion meeting the requirements of RECIST version 1.1; If the focus that has previously received local treatment (radiotherapy, ablation, vascular intervention, etc.) is the only focus, there must be a clear imaging basis for the disease progression of the focus;
6. The ECoG score was 0 or 1;
7. The laboratory test results within 7 days before the first acceptance of the study drug must meet the following criteria:

1) Neutrophil count ≥ 1.5 × 109 / L, platelet count ≥ 100 × 109 / L, hemoglobin ≥ 90 g / L (no blood transfusion, no blood products, no granulocyte colony stimulating factor or other hematopoietic stimulating factors within 7 days before laboratory examination);

2) Total serum bilirubin ≤ 1.5 × Upper normal value (ULN);

3) In the absence of liver metastasis, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 1.5 × ULN； ALT and AST ≤ 3 in patients with liver metastasis or liver cancer × ULN；［ Asymptomatic mild and moderate liver injury (defined as NCI CTCAE grade 1 toxicity) and elevated ALT and AST > 5 ~ 20 × Patients with ULN (NCI CTCAE Level 3) may tolerate the same dose of study drugs as patients with normal liver function. Patients with mild to moderate liver injury can be included on the premise that non clinical and clinical data (including pharmacokinetic and pharmacokinetic results) suggest that there is no unreasonable risk. If it is necessary to include patients with severe liver injury, it is necessary to discuss with the regulatory authority]

4) Serum creatinine ≤ 1.5 × ULN and creatinine clearance ≥ 60 ml / min (calculated according to Cockcroft Gault formula);

5) Urine routine examination showed that urinary protein was < 2 +; If urinary protein ≥ 2 +, 24-hour urinary protein quantification should be < 1 g;

6) International normalized ratio (INR) ≤ 1.5 and partially activated prothrombin time (APTT) ≤ 1.5 × ULN。

8. Expected survival ≥ 12 weeks;

9. Agree to abide by the regulations on smoking, drinking, diet and exercise restrictions during the study (which may cause more protocol violations, which shall be set according to the needs of the study);

10. Female subjects / patients of childbearing age or male subjects / patients whose partners are women of childbearing age shall take effective contraceptive measures, such as double barrier contraceptive methods, condoms, intrauterine devices, abstinence, etc., from at least 1 month before receiving the study drug for the first time to 6 months after receiving the study drug for the last time.

Exclusion Criteria:

Those who meet any of the following exclusion criteria must be excluded from the study:

1. The toxicity of previous anti-tumor treatment has not recovered ≤ grade 1 (except hair loss, skin pigment change or neurotoxicity ≤ grade 2);
2. Other malignant tumors in the past 5 years (except skin basal cell carcinoma or squamous cell carcinoma and cervical carcinoma in situ that have been effectively controlled); (according to FDA guideline 1, patients with the same or different tumor types who have been or are currently complicated with the same or different tumor types, whose medical history or treatment has no potential impact on the safety or efficacy evaluation of the study drug, should be included in the clinical study. For example, patients with previous or current malignant tumors should not be excluded in dose exploration, preliminary efficacy evaluation or proof of concept study)
3. There was central nervous system (CNS) metastasis in the past or screening, but the primary central solitary fibrous tumor can be included in the group;
4. Have received approved systemic anti-tumor therapy within 4 weeks before receiving the study drug for the first time, including chemotherapy (chemotherapy, biotherapy, targeted therapy (the washout period of small molecule targeted drugs is 2 weeks or 5 half lives, whichever is shorter), hormone therapy and traditional Chinese medicine therapy (for traditional Chinese medicine therapy with clear anti-tumor indications in the instructions, it can be treated after 1 week washout period before the first medication) Etc;
5. Radical radiotherapy (including more than 25% bone marrow radiotherapy) within 4 weeks before receiving the study drug for the first time; brachytherapy (such as implantation of radioactive particles) within 60 days before receiving the study drug for the first time; palliative radiotherapy for bone metastases within 1 week before receiving the study drug for the first time;
6. Major surgery (the definition of major surgery refers to grade 3 and 4 operations specified in the measures for the administration of clinical application of medical technology implemented on May 1, 2009) or unhealed wounds, ulcers and fractures within 4 weeks before receiving the study drug for the first time;
7. Prohibited combination drugs were used within 1 week before the first acceptance of the study drug or within 5 drug half-life (whichever is longer)
8. Within the first 4 weeks of the first study, any live vaccine or attenuated vaccine will be inoculated during the study period.
9. Previously received anti-angiogenic TKI drugs;
10. At present, there is uncontrolled malignant pleural effusion, ascites or pericardial effusion (defined as that it cannot be effectively controlled by diuretics or puncture according to the judgment of the researcher);
11. Gastrointestinal diseases such as gastric and duodenal active ulcer and ulcerative colitis, or active bleeding of unresected tumors, or other conditions that may cause gastrointestinal bleeding and perforation determined by the researcher before the study;
12. Patients with evidence or history of thrombosis or obvious bleeding tendency within 2 months before receiving the study drug for the first time (bleeding > 30 ml within 2 months, hematemesis, black stool and bloody stool), hemoptysis (fresh blood > 5 ml within 4 weeks);
13. Arterial thrombosis or deep venous thrombosis occurred within 6 months before the first study drug; or thromboembolic events (including stroke events and / or transient ischemic attack) occurred within 12 months;
14. Have active pulmonary tuberculosis, are receiving anti tuberculosis treatment or have received anti tuberculosis treatment within 1 year before receiving the study drug for the first time;
15. Patients with previous and current history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, severe impairment of lung function and other patients who may interfere with the detection and treatment of suspected drug-related pulmonary toxicity; radiation pneumonia in radiotherapy area is allowed;
16. Hepatitis B virus (HBV) DNA>1 is known to have clinically significant liver disease history, including viral hepatitis active infection (hepatitis B surface antigen HBsAg) and / or hepatitis B core antibody (HBcAb) positive. × 103 copies / ml or > 2000 IU / ml; Hepatitis C virus (HCV) antibody is known to be positive and HCV RNA > 1 × 103 copies / ml], or other hepatitis, clinically significant moderate and severe liver cirrhosis;
17. Human immunodeficiency virus (HIV) antibody positive;
18. Meet any of the following criteria related to cardiac function:

    * Various clinically significant arrhythmias or conduction abnormalities require clinical intervention;
    * At rest, the QT interval (QTCF) of electrocardiogram (ECG) was > 480 msec;

    Note: if ECG cannot directly display QTCF results, please use the following formula for calculation: QTCF = QT / ∛ RR

    • Various clinically significant cardiovascular diseases, including acute myocardial infarction, severe or unstable angina pectoris, coronary artery bypass grafting, New York Heart Function Classification (NYHA) III / IV congestive heart failure, ventricular arrhythmia requiring treatment, or left ventricular ejection fraction (LVEF) < 50% within 6 months before the first study.
19. Women who are known to be pregnant or breastfeeding;
20. Known history of allergy to the relevant components of the study drug;
21. Subjects / patients who participated in other intervention clinical studies within 4 weeks before the first acceptance of the study drug;
22. There is any disease or condition affecting drug absorption, or the subject / patient cannot take the drug orally;
23. Those who have a history of psychotropic substance abuse and cannot quit or have mental disorders;
24. For other reasons, the researcher judged that it was not suitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2021-11-21 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
PFS | 2 months
  progression free survival

SECONDARY OUTCOMES:
ORR | 2 months
  objective response rat
OS | 6 months
  over survival
DCR | 2 months
  disease control rate
DoR | 2 months
  duration of response
TTR | 2 months
  time to response
AE | 2 months
  Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Xiaowei Zhang, Doctor, Study Chair — Fudan Cancer Center，Shanghai
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided